CLINICAL TRIAL: NCT07052734
Title: A Multicenter Retrospective Analysis of the Miti-gene Recurrence Score in Early-Stage Invasive HR-Positive, HER2-Negative Breast Cancer in China
Brief Title: Miti-gene Recurrence Score in HR+/HER2- Chinese Breast Cancer Patients
Acronym: BC-MRS-01
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wang shusen, Professor, Sun Yat-sen University
Other Study IDs: BC-MRS-01
Record Dates: First submitted 2025-06-28; First posted 2025-07-06 (Actual); Last update posted 2025-07-06 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Update and validate the performance of the 21-gene score in prognostic stratification for early-stage HR-positive, HER2-negative breast cancer in China.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed age: 18-75 years.
2. Early-stage invasive breast cancer, pN0-1.
3. Molecular subtype: HR-positive (ER and/or PR positive), HER2-negative.
4. At least five years of follow-up records (including cases with disease progression within five years and documented records).
5. Sufficient FFPE samples for sectioning or frozen samples for RNA extraction and subsequent testing.

Exclusion Criteria:

1. FFPE samples with tumor content <20%, and inability to enrich tumor regions through cutting.
2. Insufficient extracted nucleic acid quantity or severe degradation preventing further experiments.
3. Failure in RT-PCR amplification of housekeeping genes.
4. Multiple primary breast cancers or a history of ipsilateral or contralateral breast cancer.
5. Disease progression unrelated to breast cancer.
6. Lack of prior signed consent for retrospective scientific research or exemption from informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR-positive, HER2-negative breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 2843 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 10 years
  Disease-Free Survival (DFS) is defined as the duration from the completion of curative surgery until the first occurrence of any of the following events: local or distant relapse of the breast cancer, development of a new primary cancer, or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 10 years
  Overall survival is defined as the duration from the completion of curative surgery until death from any cause.
Distant relapse-free survival | 10 years
  Distant relapse-free survival is defined as the duration from the completion of curative surgery until distant relapse of the breast cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China